CLINICAL TRIAL: NCT03988101
Title: Role of Statin in Venous Dysfunction in Patients With Venous Thromboembolism Event
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2018-0726
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Venous Thromboembolism; Dyslipidemias
MeSH Terms: conditions — Venous Thromboembolism; Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: A prospective placebo-controlled, double-blind, phase IV clinical study to evaluate the efficacy and safety of statin in patient with venous dysfunction
Who Masked: Participant, Care Provider, Investigator
Masking Description: Researchers, research coordinators, and subjects are all blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin 20mg (Experimental): Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of rosuvastatin 20 mg once daily or equivalent.
  Interventions: Drug: Rosuvastatin 20mg
- Control (Placebo Comparator): Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of rosuvastatin 20 mg once daily or equivalent.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Rosuvastatin 20mg — Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of rosuvastatin 20 mg once daily or equivalent.
  Arms: Rosuvastatin 20mg
Drug: Control — Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of rosuvastatin 20 mg once daily or equivalent.
  Arms: Control

SUMMARY:
Participants between the ages of 19 and 70 who were initially diagnosed with venous thromboembolism and were accompanied by dyslipidemia (LDL> = 100 mg / dl) were enrolled.

Participants diagnosed with pulmonary embolism, pulmonary embolism CT, and peripheral B-mode ultrasound (B-mode ultrasound) Only participants who do not meet the exclusion criteria should be enrolled in the study.

Once the participant is selected, the patient is informed of the study and receives the consent form.

Participants who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of rosuvastatin 20 mg once daily or equivalent. Participants who previously used statins have a wash-out period of two weeks or more Participants undergo a visit at 12 weeks after initiation of treatment. For fasting blood tests, patients visit on an empty stomach. Outpatient follow-up observes side effects after last visit and observes changes in vital signs and weight.

After 24 weeks of treatment, the participant visits for efficacy evaluation. We performed body weight, vital signs and blood tests (WBC, hemoglobin, BUN, creatinine, CRP, D-dimer, fibrinogen, PAI-1, AST, ALT, CK, total cholesterol, triglyceride, HDL and LDL).

1. Primary evaluation item: Improvement of venous insufficiency at 6 months
2. Secondary evaluation items: Improvement of blood lipid concentration, inflammation and blood clotting at 6 months Comparison of numerical rate of change
3. Tertiary evaluation items: recurrence of venous thrombosis

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who were initially diagnosed with venous thromboembolism
* 2. Patients who were between 19 and 70 years of age with dyslipidemia (LDL> = 100 mg / dl)

Exclusion Criteria:

* 1. Under 18
* 2. Active cancer status
* 3. Known CVD (ischemic heart disease, stroke, peripheral artery disease)
* 4. LDL> 190ml / dL or LDL <100mg / dL
* 5. Contraindication for anticoagulation (NOAC)
* 6. Contraindication for Statin(Pregnancy, Breastfeeding, Active liver disease, Elevation of liver enzymes, Allergic reaction to a statin)
* 7. Patients with vital sign unstable with Massive VTE
* 8. DVT remains in the vascular ultrasound

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
The improvement rate of venous insufficiency | 6months
  Venous function test (test items according to research) - DVT doppler(thrombus, spontaneous echo contrasts, compressibility)
The improvement rate of venous insufficiency | 6months
  Venous function test (test items according to research) - Venous insufficiency doppler (reflux, reflux site)

SECONDARY OUTCOMES:
Comparison of changes in lab data | 6months
  Comparison of changes in blood lipid levels, inflammation, and blood coagulation
  - Test items according to standard treatment WBC, Hemoglobin, BUN, Creatinine, CRP, D-dimer, Fibrinogen, PAI-1
Comparison of changes in lab data | 6months
  Comparison of changes in blood lipid levels, inflammation, and blood coagulation
  - Test items according to research AST, ALT, CK, total cholesterol, triglyceride, HDL, LDL

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
When you request the material you want, I can consider giving the requested material.
  If you have any questions, please contact grhong@yuhs.ac